CLINICAL TRIAL: NCT04948346
Title: Relationship Between N-trimethylamine Oxide, a Metabolite of Intestinal Flora, and Pathogenesis and Progression of Amyotrophic Lateral Sclerosis
Brief Title: Correlation Between Intestinal Microflora Metabolites and Amyotrophic Lateral Sclerosis
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2017358
Record Dates: First submitted 2021-06-27; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient with ALS
  Interventions: Other: diagnosed with ALS
- patient'spouse(without ALS)

INTERVENTIONS:
Other: diagnosed with ALS — diagnosed with ALS
  Groups: patient with ALS

SUMMARY:
To verify the correlation between TMAO level and the pathogenesis and progression of ALS

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a fatal neurodegenerative disease with rapid progression, poor prognosis and unknown etiology. At present, there is no effective treatment. In recent years, with the deepening of the research on the interaction between intestinal flora and human health, many studies have found that intestinal flora is closely related to neurodegenerative diseases. In the field of neuroscience, there are more and more researches on the relationship between TMAO and its precursors (L-carnitine, etc.) and neurodegenerative diseases. Although there is no direct study on the relationship between TMAO and ALS, the relevant experiments suggest that intestinal flora, TMAO and its precursors (L-carnitine, etc.) may be involved in the pathogenesis and progression of ALS. The purpose of this study is to verify the important role of TMAO, a metabolite of intestinal flora, in ALS through human studies and animal model studies, and to obtain direct evidence that TMAO participates in the disease process of ALS.

ELIGIBILITY:
Inclusion Criteria:

* ① ALS patients in outpatient or ward voluntarily participated in the study and signed informed consent by themselves or their authorized family members; ② At the time of enrollment, the diagnostic grade of ALS patients met the criteria of the World Federation of Neurology (WFN) revised in 1998; ③ They were 18-75 years old; ④ Antibiotics, L-carnitine and intestinal flora regulation were not used within 3 months; ⑤ Can eat normally.

Exclusion Criteria:

* ① electromyography detection found motor nerve block, sensory nerve conduction abnormalities, or imaging examination (CT or MRI) found lesions that could explain the clinical manifestations of patients, which did not support the diagnosis of ALS; ② The patients with dementia or mental disorder could not cooperate with the researchers; ③ Patients with severe heart, liver, kidney and other severe concomitant diseases; ④ Patients with gastrointestinal diseases or gastrointestinal surgery may affect gastrointestinal absorption; ⑤ The patients who were treated with antibiotics, L-carnitine and intestinal flora regulation in recent 3 months; ⑥ Breast feeding or pregnancy; ⑦ Patients with dysphagia, inability to eat normal food, or indwelling gastric tube or gastrostomy for enteral nutrition.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with Sporadic ALS
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Plasma TMAO levels | 6 month after inclusion into the study
  Plasma TMAO levels in ALS patients and their spouses

SECONDARY OUTCOMES:
Change rate of frs-r score | 6 month after inclusion into the study
  Change rate of frs-r score in ALS patients

CONTACTS AND LOCATIONS:
Overall Officials: Lu Chen, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No